CLINICAL TRIAL: NCT01950975
Title: Screening for Chromosomal Microarrangements by CGH-array in Developmental Anomalies of the Skin Suggestive of Mosaicism. National Multicentre Descriptive Study.
Brief Title: Screening for Chromosomal Microarrangements by CGH-array in Developmental Anomalies of the Skin Suggestive of Mosaicism.
Acronym: MOSAÏQUE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: VABRES PHRC N 2010
Record Dates: First submitted 2013-08-27; First posted 2013-09-26 (Estimated); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Malformations With Skin Manifestations Suggesting Mosaicism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Parents (Other): 2 parents of child
  Interventions: Biological: Peripheral blood samples in EDTA tubes
- infant (Other)
  Interventions: Biological: Peripheral blood samples in EDTA tubes; Procedure: Skin biopsies

INTERVENTIONS:
Biological: Peripheral blood samples in EDTA tubes
Procedure: Skin biopsies
  Arms: infant

SUMMARY:
The principal result expected is the discovery of inframicroscopic chromosomal rearrangements in regions of the genome not yet known to be involved, or mutations in known candidate genes;

The identification of such a mosaic rearrangement in an affected infant would lead to improved genetic counselling. Indeed, as this mosaicism is a consequence of a genetic event occurring at an early stage of embryogenesis, it would be possible to confirm the sporadic nature of the observed disorder and therefore to predict a very low or even negligible risk of recurrence for the couple concerned. For the affected infant, the risk for his/her own offspring will be assessed according to the nature of the genetic anomaly discovered. For medical practice, investigators hope that this study will lead to a clearer definition of the screening modalities for mosaicism in the disorders concerned. In particular, they hope to determine whether or not it is possible to dispense with a skin biopsy, which is more invasive than a blood sample.

ELIGIBILITY:
Inclusion Criteria:

* Persons who have provided written informed consent
* Lower age limit: infant born at more than 37 WA
* Sporadic disorder
* Patients presenting at least two skin criteria, or one skin criterion and one non-skin criterion
* Skin criteria: 1- extensive epidermal or sebaceous naevus, 2- Extensive "segmental" haemangioma, 3- Flat angioma or extensive complex vascular malformation, 4-Pigmentary disorders with patterns suggesting mosaicism (Blaschko lines)
* Non-skin criteria: Cerebral, ocular, cardiac or genito-urinary malformation, asymmetric body, segmental hypertrophy of a limb, spinal dysraphism (only when associated with haemangioma)

Exclusion Criteria:

* Persons not covered by the national health insurance scheme
* Mendelian disorders: CM-AVM syndrome, glomangiomatosis, Cowden or Bannayan syndrome, type 1 neurofibromatosis, incontinentia pigmenti, CHILD syndrome, Happle-type chondrodysplasia punctata
* Mendelian mosaic disorders: epidermal or epidermolytic, comedo or dyskeratotic nevus.
* Family history of one of these disorders
* Suspicion or an autosomal dominant disease
* Patient and/or parent under guardianship or ward of court

Min Age: 37 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 315 (Actual)
Dates: Start 2012-02-20 (Actual); Primary Completion 2017-09-08 (Actual)

PRIMARY OUTCOMES:
Presence or not of inframicroscopic chromosomal rearrangements | baselines

SECONDARY OUTCOMES:
Rate of detection of a chromosomal anomaly | baselines

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Dijon, Dijon, France

REFERENCES:
- [Derived] Faivre L, Crepin JC, Reda M, Nambot S, Carmignac V, Abadie C, Mirault T, Faure-Conter C, Mazereeuw-Hautier J, Maza A, Puzenat E, Collonge-Rame MA, Bursztejn AC, Philippe C, Thauvin-Robinet C, Chevarin M, Abasq-Thomas C, Amiel J, Arpin S, Barbarot S, Baujat G, Bessis D, Bourrat E, Boute O, Chassaing N, Coubes C, Demeer B, Edery P, El Chehadeh S, Goldenberg A, Hadj-Rabia S, Haye D, Isidor B, Jacquemont ML, Van Kien PK, Lacombe D, Lehalle D, Lambert L, Martin L, Maruani A, Morice-Picard F, Petit F, Phan A, Pinson L, Rossi M, Touraine R, Vanlerberghe C, Vincent M, Vincent-Delorme C, Whalen S, Willems M, Marle N, Verkarre V, Devalland C, Devouassoux-Shisheboran M, Abad M, Rioux-Leclercq N, Bonniaud B, Duffourd Y, Martel J, Binquet C, Kuentz P, Vabres P. Low risk of embryonic and other cancers in PIK3CA-related overgrowth spectrum: Impact on screening recommendations. Clin Genet. 2023 Nov;104(5):554-563. doi: 10.1111/cge.14410. Epub 2023 Aug 14. PMID 37580112
- [Derived] Sorlin A, Maruani A, Aubriot-Lorton MH, Kuentz P, Duffourd Y, Teysseire S, Carmignac V, St-Onge J, Chevarin M, Jouan T, Thauvin-Robinet C, Thevenon J, Faivre L, Riviere JB, Vabres P. Mosaicism for a KITLG Mutation in Linear and Whorled Nevoid Hypermelanosis. J Invest Dermatol. 2017 Jul;137(7):1575-1578. doi: 10.1016/j.jid.2017.01.035. Epub 2017 Feb 28. No abstract available. PMID 28257793